CLINICAL TRIAL: NCT07164755
Title: Measurement of Serum Cytokine Levels in Samples Collected as Part of a Clinical Trial of Psilocybin for Treatment-resistant Depression.
Brief Title: Measurement of Serum Inflammatory Markers in Patients Treatment-resistant Depression Given Psilocybin
Status: Active, not recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 357453
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psilocybin-treated group blood samples: Blood samples from participants in Psider trial treated with psilocybin 25mg
- Placebo-treated group blood samples: Blood samples from participants in Psider trial treated with placebo

SUMMARY:
About one in three people with major depression respond poorly to standard antidepressant treatments. This kind of depression is called treatment-resistant depression, and it can lead to long-term disability, financial challenges, and a higher risk of suicide.

Psilocybin-a compound found in certain mushrooms-has shown early promise as a new treatment for this difficult-to-treat depression. Scientists believe it works by affecting a specific brain receptor (called 5-HT2A), which helps the brain become more flexible and adaptable. But there's another possible mechanism of psilocybin that hasn't been studied much: its ability to influence the immune system.

Recent research suggests that inflammation in the body might play a role in depression, especially when treatments don't work. High levels of certain inflammatory markers (called cytokines) are linked to poor response to antidepressants, while lower levels are tied to feeling better. Psilocybin may help reduce this inflammation, which could be part of why it helps some people feel better.

Still, we don't fully understand how a person's inflammation levels before treatment, and how those levels change afterward, relate to how well psilocybin works. Figuring this out could help doctors better match patients to psychedelic therapy and discover new ways to treat depression.

In this study, blood samples from a recent study (called the PsiDeR trial) that tested psilocybin in people with treatment-resistant depression will be analyzed. Cytokine levels in these blood samples, as well as levels of another type of molecule linked to inflammation, called mRNA, will be measured.

DETAILED DESCRIPTION:
Chronic and elevated inflammation is associated with depression. Depressed patients tend to have raised inflammatory markers compared to healthy controls, and studies have reported that the greatest elevation is seen in patients with treatment-resistant depression (TRD). Previous studies highlight the bidirectional relationship between inflammation and depression. Elevated pro-inflammatory cytokines are linked to poor antidepressant response, while reductions in these markers are associated with symptom improvement. While neuroinflammation may play a role in the pathophysiology of depression, inflammation is also a causal risk factor for physical illnesses that are often co-morbid with depression, such as cardiovascular disease. As such, targeting inflammation in patients with depression may have significant implications for both their mental and physical health.

Psychedelics are emerging as a potential new class of therapeutic agents for psychiatric illness, including depression. It has been suggested that their therapeutic effect may partly be due to reducing inflammation. Psychedelics have been shown reduce markers of inflammation in models of human inflammatory disease, both in vitro and in vivo. While, as might be expected, psilocybin was not found to reduce markers of inflammation in healthy human volunteers, in a clinical sample of people with treatment-resistant depression, use of ayahuasca (containing the psychedelic N,N DMT) resulted in a significant reduction in CRP levels compared to participants given placebo, with the reduction in CRP levels significantly correlated with a reduction in depressive symptoms. Ayahuasca consists of an admixture of multiple different compounds. As such, the relative contribution of the psychedelic to the anti-inflammatory effect that was observed is unknown.

The effect of isolated psychedelic compounds such as psilocybin on the systemic inflammatory state of patients, specifically patients with depression, therefore, remains to be investigated. Psilocybin's capacity to reduce inflammation, as evidenced in preclinical models, may be a crucial mechanism underlying its therapeutic effects. Moreover, while it is recognised that baseline inflammation levels can influence the effectiveness of conventional antidepressants, it is unclear whether this is also the case for psilocybin.

This study aims to evaluate serum cytokine and inflammatory-related mRNA levels in samples collected from participants with TRD who took part in the (Psi)locybin in (De)pression (R)esistant to Standard Treatments (PsiDeR) Trial, and the relationships between these and psilocybin treatment response. PsiDeR was a randomised, placebo-controlled trial of psilocybin as a treatment for TRD that has now completed.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in the English language
* Fulfil Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5) criteria for current single or recurrent episodes of MDD of at least moderate severity but without psychotic features, as defined on the MINI 7.0.
* 17-item HAM-D score ≥ 14.
* Have failed to respond to 2 or more antidepressants prescribed at the minimum effective dose for at least 6 weeks OR at least 1 antidepressant prescribed at the minimum effective dose for at least 6 weeks AND a course of evidence-based psychotherapy given for at least 6 sessions.
* For those aged ≥ 60 years, the first episode of depression must have started prior to their 60th birthday.

Exclusion Criteria:

Diagnosis of bipolar disorder (defined as meeting DSM-5 criteria for bipolar 1 or bipolar 2) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.

Diagnosis of psychotic disorder (defined as meeting DSM-5 criteria for any psychotic disorder) on the MINI 7.0, EXCEPT substance/medication induced psychotic disorder where the duration was limited to the acute period of direct intoxication with the substance/medication. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.

Diagnosis of drug or alcohol dependence syndrome (defined as meeting DSM-5 criteria for any dependence syndrome) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.

Diagnosis of any personality disorder (defined as meeting DSM-5 criteria for any personality disorder) based on clinical interview and the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.

Diagnosis of any dementia (defined as meeting DSM-5 criteria for any dementia disorder) based on clinical interview by a psychiatrist.

Personal history of a ≥ 1 suicide attempt in the past year requiring hospitalization, defined using the CSSRS (Q6 (past year) = "y") and confirmation at clinical interview with a psychiatrist.

Other personal circumstances and behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin.

Depression secondary to other medical conditions

Medical diagnosis incompatible with psilocybin treatment

Inability to provide a screening blood sample, urine sample or electrocardiogram.

Biochemical abnormalities (defined as falling outside the normal reference range) as evaluated by a full blood count, full biochemistry profile and thyroid function tests. Biochemical abnormalities must also be determined as clinically significant by a medical doctor to fulfil the criterion for exclusion.

Electrocardiographic abnormalities, defined as any abnormality that is not normal sinus rhythm and determined as clinically significant by a medical doctor.

Women of child bearing potential not using adequate contraception.

Pregnant or breast-feeding women.

Those unable to give informed consent.

Non-registration with a GP or failure to consent to sharing of the GP summary care record and any psychiatric assessments held.

Those enrolled in another drug trial

Hypersensitivity to the IMP or to any of the excipients or placebo

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment-resistant depression, recruited in the UK
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Linear regression to examine the association between baseline cytokines and depression outcomes at six weeks | Six weeks
  Linear regression to examine the association between baseline cytokines and depression outcomes at six weeks

SECONDARY OUTCOMES:
Linear regression to examine the association between cytokine level change and depression outcomes at six weeks. | Six weeks
  Linear regression to examine the association between cytokine level change and depression outcomes at six weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided